CLINICAL TRIAL: NCT01069731
Title: Comparison of NNS Performance Measures to Clinical Estimates of Suck and Feeding Readiness in Preterm Infants Using the NTrainer Device
Brief Title: Comparison of Non-nutritive Suck (NNS) Measures to Clinical Estimates of Suck and Feeding Readiness in Preterm Infants
Status: Completed | Type: Observational
Sponsor: KC BioMediX, Inc (Industry)
Responsible Party: Thomas Young, MD, WakeMEd
Other Study IDs: WakeMed Study 748
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Preterm Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Infants born at 30 to 36 weeks gestation: Infants will be considered eligible if they are born at 30 to 36 weeks gestation and have no exclusion criteria.

SUMMARY:
This is a research study to quantitatively assess the development of non-nutritive suck (NNS) and feeding readiness in preterm infants using a novel device, the NTrainer©, and to compare this with two clinical assessment tools, NOMAS and EFS.

DETAILED DESCRIPTION:
Fifteen minutes before feeding, the mobile NTrainer recording station will be positioned cribside. Following a brief exam of physiologic state, using the Oral Feeding Readiness Assessment portion of the EFS, the infant will be cradled in a supportive inclined posture, swaddled, with limbs positioned at midline, and background/overhead lighting dimmed in the area to promote eye contact with the tester. Sampling of NNS behavior will not be initiated until the infant is in an optimal behavioral state, i.e., drowsy to active alert (state 3 or 4 or 5 as described by the Naturalistic Observation of Newborn Behavior, Newborn Individualized Developmental Care and Assessment Program; NIDCAP). The infant will be presented with the NTrainer pacifier, and several contiguous 30-second blocks of NNS nipple compression data will be sampled using the NeoSuck RT software. The infant will remain connected to the usual NICU monitors at all times for observation of respiration, heartbeat and oxygen saturation.

After the NTrainer data collection is completed, the baby will be fed by his or her nurse or parents as directed in the care plan. If the baby is able to feed by mouth, one of the investigators will observe the feeding, and perform 1) a NOMAS evaluation during the first 2 minutes of the feeding, and 2) an EFS assessment after the feeding is completed.

Infants will be studied in 2 sessions each day beginning at Day 4 to 7 of life, then twice weekly (2 sessions per day, 2 days per week) until hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Born at 30 to 36 weeks gestation and have no exclusion criteria.

Exclusion Criteria:

* Significant birth defects.
* Breathing difficulties severe enough to require being on a ventilator or nasal CPAP for more than 2 hours after birth.
* Any oxygen requirement at Day 4 of life.
* Any neurologic problems, including seizures or frequent apnea spells.

Ages: 30 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants born prematurely may suffer multiple adverse events in the NICU, and these experiences may negatively impact normal developmental processes of immature cardiorespiratory, gastrointestinal and central nervous systems. As a result, many infants have at least transient difficulties learning to successfully manage oral feedings. Oral feeding difficulties in the NICU may prolong the time to discharge, cause significant parental anxiety, and persist throughout infancy.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To describe NNS pressure waveforms and NNS-STI values in normal premature infants with gestational ages 30 to 36 weeks during the first week of life. | First Weeks of Life

SECONDARY OUTCOMES:
To describe the progression of NNS waveform pattern and NNS-STI values in normal premature infants as they mature to term postmenstrual age. | Mature to full term postmenstrual age

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Young, MD, Principal Investigator — WakeMed Health and Hospitals
Locations (1):
- WakeMed, Raleigh, North Carolina, United States

REFERENCES:
- [Background] Barlow SM, Finan DS, Lee J, Chu S. Synthetic orocutaneous stimulation entrains preterm infants with feeding difficulties to suck. J Perinatol. 2008 Aug;28(8):541-8. doi: 10.1038/jp.2008.57. Epub 2008 Jun 12. PMID 18548084